CLINICAL TRIAL: NCT01893242
Title: A PHASE III RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE POTENTIAL OF ALEGLITAZAR TO REDUCE THE RISK OF END STAGE RENAL DISEASE AND CARDIOVASCULAR MORTALITY IN PATIENTS WITH TYPE 2 DIABETES AND CHRONIC KIDNEY DISEASE (ALERENAL STUDY)
Brief Title: A Study of Alegitazar in Patients With Type 2 Diabetes And Chronic Kidney Disease (Alerenal Study)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC28504; 2013-000088-10 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2, Kidney Disease, Chronic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases; Bronchiolitis Obliterans Syndrome | interventions — aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar Arm (Experimental)
  Interventions: Drug: Aleglitazar
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aleglitazar — Aleglitazar 150 mcg oral doses, once a day for approximately 3 years
  Arms: Aleglitazar Arm
Drug: Placebo — Matching placebo to aleglitazar, once a day for approximately 3 years
  Arms: Placebo Arm

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the potential of aleglitazar to reduce the risk of end stage renal disease and cardiovascular mortality in patients with type 2 diabetes mellitus and chronic kidney disease. Patients will be randomized to receive oral daily doses of aleglitazar or matching placebo. The anticipated time on study treatment is approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 18 years of age at screening
* Diagnosis of diabetes mellitus Type 2
* Glycosylated hemoglobin A1C (HbA1C) < 10% at screening
* Estimated glomerular filtration rate (eGFR) >=30 and < 60 mL/min/1.73 m2
* Urinary albumin-to-creatinine ratio (UACR) >=500 and < 5000 mg/g
* Treatment with either angiotensin converting enzyme inhibitor or angiotensin II receptor blocker for at least three months prior to screening
* Women of child-bearing potential using a highly effective birth control method must be willing to use the same method of contraception during the entire course of the study

Exclusion Criteria:

* Treatment with a PPARgamma agonist and/or PPARalpha agonist in the last 12 weeks screening
* Prior intolerance to a TDZ or fibrate
* Previous participation in a trial with aleglitazar
* Diagnosis or history of other types of diabetes
* Diagnosis or history of acute metabolic diabetic complications within the past 6 months
* Known primary glomerulonephritis, secondary glomerulonephritis other than diabetic nephropathy or polycystic kidney disease
* Diagnosed acute kidney injury or dialysis within 12 weeks prior to screening
* Poorly controlled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg at baseline)
* Known secondary hypertension due to renal artery stenosis, primary aldosteronism, or pheochromocytoma
* History of myocardial infarction or stroke in the past 12 weeks prior to screening
* Symptomatic congestive heart failure NYHA class II-IV at baseline or heart failure leading to hospitalization within the 12 months prior to screening
* Diagnosed and/or treated malignancy (except for treated cases of basal cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) within the past 5 years
* Inadequate liver and hematological function
* Chronic treatment with immunosuppressive therapy
* Women who are pregnant, intending to become pregnant during the study period, currently lactating females, or women of child-bearing potential not using highly effective birth control methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of either component of the composite endpoint: end stage renal disease or cardiovascular death | Approximately 5 years

SECONDARY OUTCOMES:
Time to the first occurrence of any component of major adverse cardiovascular event composite (cardiovascular death, non-fatal myocardial infarction, non-fatal stroke) | Approximately 5 years
Time to the first occurrence of any component of macrovascular composite (CV death, non fatal myocardial infarction, hospitalization for unstable angina, non fatal stroke) | Approximately 5 years
Time to the first occurrence of any component of composite outcome of end-stage renal disease and all-cause mortality | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche